CLINICAL TRIAL: NCT03172468
Title: Definition of Hemodynamic Thresholds in Out-of-Hospital Cardiac Arrest: Advancing Advanced Life Support Towards Goal Directed Resuscitation
Brief Title: Definition of Hemodynamic Thresholds in Out-of-Hospital Cardiac Arrest
Acronym: HETOCA
Status: Withdrawn | Type: Observational
Why Stopped: unable to facilitate patient recruitment
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HETOCA-2017-v1.1
Record Dates: First submitted 2017-05-15; First posted 2017-06-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients suffering from out-of-hospital cardiac arrest (OHCA), who achieve sustained return of spontaneous circulation (ROSC) following prehospital cardiopulmonary resuscitation.
- Non-Survivors: Patients suffering from out-of-hospital cardiac arrest (OHCA), who are declared dead after prehospital cardiopulmonary resuscitation.

SUMMARY:
This study seeks to evaluate, whether patients suffering from cardiac arrest, that can be successfully resuscitated, can be differentiated from those, that cannot be resuscitated, using arterial blood pressure values.

DETAILED DESCRIPTION:
Cardiopulmonary resuscitation (CPR) in patients suffering from cardiac arrest out of hospitals is based on strict clinical practice guidelines. However, the evidence base for these treatment recommendation is insufficient in many respects. While knowledge about basic interventions, that are capable of restoring spontaneous circulation and improving neurologically intact survival - chest compressions, application of oxygen and early defibrillation -, has increased over the last decade, advanced treatment options - advanced airway management, vascular access, application of vasoactive drugs - are still recommended, although clinical trials of varying quality failed to demonstrate any benefit in patient related outcomes.

This study seeks to establish hemodynamic threshold values that are able to discriminate between patients that achieve return of spontaneous circulation (survivors) and those that fail to do so (non-survivors). These cutoff values could act as targets for interventions during CPR (i.e. application of vasoactive drugs, use of mechanical compression devices, …) in further trials and may potentially influence clinical practice later on. Furthermore, reliable cutoff values could act as additional prognostic factors during CPR, enabling prehospital care providers to base their decisions to continue or terminate ongoing CPR efforts on a more solid basis.

To achieve this goal, 22 patients with out-of-hospital cardiac arrest (OHCA) treated by physicians of the prehospital physician response system located at the Medical University of Graz shall be included into this trial. All patients will receive Advanced Life Support (ALS) interventions according to current guidelines issued by the European Resuscitation Council (ERC). In addition, arterial lines will be placed and arterial blood pressure will be measured continuously. This intervention is already considered standard of care at this prehospital physician response system and performed routinely as part of the local ALS algorithm.

Relevant parameters - systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP) etc. - will be documented electronically using both the electronic documentation system already used by the prehospital physician response system and the monitor/defibrillator device. Median values will be compared between survivors and non-survivors and possible threshold values will be calculated. Cutoff values that would be best suited to act as targets in future research and clinical practice will be identified by receiver operating characteristics (ROC).

ELIGIBILITY:
Inclusion Criteria

* Out-of-hospital cardiac arrest
* Age >18 years
* Advanced Life Support started
* Arterial line placement possible

Exclusion Criteria

* Obvious signs of death
* Advanced Directives / Do Not Attempt Resuscitation Order
* Cardiac arrest of traumatic etiology
* Documented patient refusal in advance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from cardiac arrest on arrival of the physician response unit are to be included, if ALS is deemed reasonable by the emergency physician. The groups to be compared are survivors (patients with sustained return of spontaneous circulation (ROSC) in the field who are transported to a hospital alive) and non-survivors (patients in whom CPR is terminated in the field).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Blood Pressure | immediately after placement of the arterial line
  Mean arterial blood pressure measured invasively via the arterial line.

SECONDARY OUTCOMES:
Systolic Arterial Blood Pressure | immediately after placement of the arterial line
  Systolic arterial blood pressure measured invasively via the arterial line.
Diastolic Arterial Blood Pressure | immediately after placement of the arterial line
  Diastolic arterial blood pressure measured invasively via the arterial line.
Mean Arterial Blood Pressure | one minute after the first application of epinephrine following placement of the arterial line
  Mean arterial blood pressure measured invasively via the arterial line.
Systolic Arterial Blood Pressure | one minute after the first application of epinephrine following placement of the arterial line
  Systolic arterial blood pressure measured invasively via the arterial line.
Diastolic Arterial Blood Pressure | one minute after the first application of epinephrine following placement of the arterial line
  Diastolic arterial blood pressure measured invasively via the arterial line.
Mean Arterial Blood Pressure | five minutes after placement of arterial line
  Mean arterial blood pressure measured invasively via the arterial line.
Systolic Arterial Blood Pressure | five minutes after placement of arterial line
  Systolic arterial blood pressure measured invasively via the arterial line.
Diastolic Arterial Blood Pressure | five minutes after placement of arterial line
  Diastolic arterial blood pressure measured invasively via the arterial line.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Zajic, MD, Principal Investigator — Div. of General Anaesthesiology, Emergency- and Intensive Care Medicine, Medical University of Graz
Locations (1):
- Prehospital Physician Response System, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Informed Consent Form — https://box.medunigraz.at/s/QuTYym3xsqXybWI
- Available data/document: Study Protocol — https://box.medunigraz.at/s/YbufqAn3DBI1f4Q